CLINICAL TRIAL: NCT05981495
Title: Clinical Evaluation of the NanoDetect-TB Mycobacterium Tuberculosis Detection Kit for the Diagnosis of Tuberculosis Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NanoPin Technologies, Inc. (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Other Study IDs: NanoDetect-TB_01
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Extrapulmonary; Tuberculosis Active
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Extrapulmonary; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TB Suspects: TB Suspects recruited to this study will have blood drawn in a single visit.
  Interventions: Device: NanoDetect-TB

INTERVENTIONS:
Device: NanoDetect-TB — This study of the NanoDetect-TB investigational device will test plasma and serum samples from TB suspects. There is no intervention for the subjects and there will be a single visit blood draw.

SUMMARY:
The goal of this observational study is investigate the accuracy of the NanoDetect-TB kit in diagnosing tuberculosis (TB) using frozen serum and plasma samples collected from individuals suspected to have TB disease.

The main question[s] it aims to answer are:

* How does this investigational device compare to the gold standard for TB diagnosis of sputum culture?
* How does it compare to Acid-Fast Bacteria (AFB) smear microscopy and FDA-approved NAAT TB diagnostic assays?

Participants will be asked to have blood drawn and provide demographic and medical data for this study in a single visit.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults aged two years or older (including older adults that are 65+)
* Ability and willingness to provide informed consent/assent/permission, and a parent/legal guardian willing to give consent on the child's behalf for study participants aged 2-17 years
* Ability and willingness to perform study procedures, or parent/legal guardian to provide consent for a child to undergo study procedures on their behalf (when applicable)
* Clinical signs and symptoms typically associated with active TB disease including, but not limited to:

Cough for > two (2) weeks Lethargy, weakness, malaise Reduced playfulness (pediatric population) Weight loss or loss of appetite Failure to thrive (pediatric population) Fever Chest pain Night sweats

* Physician (or healthcare provider) suspicion of TB disease

Exclusion Criteria:

* Pregnancy (based on participant-provided information)
* Any physical or mental health condition for which participation in the study, as judged by the investigator, could compromise the well-being of the subject and/or prevent, limit, or confound protocol-specified procedures
* Critical illness needing immediate medical care
* Receipt of treatment for active TB or LTBI in the past 24 months

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TB suspects at clinical sites for recruitment in Houston, Miami, and New York City.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
NanoDetect-TB result compared to sputum culture | Single visit for patient for blood draw.
  The investigational device results will be compared to the primary reference of sputum culture for determining relative sensitivity and specificity.

SECONDARY OUTCOMES:
NanoDetect-TB result compared to AFB Smear and NAAT | Single visit for patient for blood draw.
  The investigational device results will be further compared to the AFB Smear and NAAT for determining relative sensitivity and specificity.

IPD SHARING:
Plan to Share IPD: No